CLINICAL TRIAL: NCT02628834
Title: Investigating the Acute Effect of Fascial Mobilization on Dynamic Walking Parameters in Patients With Multiple Sclerosis: A Crossover Controlled Group Study
Brief Title: Acute Effect of Fascial Mobilization on Gait in Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, hhotaman, PhD, PT, Hacettepe University
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D/01070
Record Dates: First submitted 2015-11-11; First posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Sclerosis
Keywords: Loading; Gait; Multiple Sclerosis; Manual Therapy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Musculoskeletal Manipulations; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fascial mobilization (Experimental): First day intervention: Patients will take fascial mobilization techniques to management of plantar flexor spasticity
  Interventions: Other: Fascial mobilization
- Stretching exercise (Experimental): Second day intervention:Patients will take fascial mobilization techniques to management of plantar flexor spasticity
  Interventions: Other: Stretching Exercise
- Healthy Volunteers (No Intervention): Healthy individuals will only be evaluated with no intervention

INTERVENTIONS:
Other: Fascial mobilization — The patient will lie on prone position with knee extension and therapist put the patient's plantar surface to her femoral region. Achilles, tibialis posterior, perenous longus and brevis distal tendons, gastrocnemius proximal tendons, hamstring's distal tendons will be mobilized at first stage. The second stage of fascia mobilization included the deep fascial mobilization of posterior crural muscle trunks. After that, the skin also will be gently mobilized. During fascial mobilization, once the spastic muscles relaxation will appeared, the ankle will move to dorsiflexion gradually. FM will carry out for 15 minutes for each foot.
  Other Names: manual therapy
  Arms: Fascial mobilization
Other: Stretching Exercise — Patients will receive also stretching exercises consisted of 30 s stretching and 10 s resting periods and will carry out for 15 minutes for each foot at second day after the first evaluation.
  Arms: Stretching exercise

SUMMARY:
Ten patients who were referred to receive physiotherapy and 10 healthy volunteers will be participants of the study.Following the initial evaluation, participants with multiple sclerosis will take the fascial mobilization for their posterior crural muscle group and hamstring distal tendons which connects the crural bones at first day. After the day following the first visit participants will asked to come again and stretching exercises will apply to plantar muscle groups after the evaluation. Every participants will evaluate with the following assessment tools: Modified Ashworth scale will use to evaluation of severity of plantar flexor spasticity. Static and dynamic loading parameters will assess with dynamic pedobarography.

DETAILED DESCRIPTION:
Ten patients who were referred to receive physiotherapy at the neurology department of Physiotherapy and Rehabilitation of the Faculty of Health Sciences of Hacettepe University, Ankara with multiple sclerosis and ten voluntary healthy age matched participants will be the subjects of this study.

Following the initial evaluation, participants with multiple sclerosis will take the fascial mobilization (FM) for their posterior crural muscle group and hamstring distal tendons which connects the crural bones at first day. After the day following the first visit participants will ask to come again and stretching exercises will apply to plantar muscle groups after the evaluation. In the investigators' study fascial mobilization will use to release plantar flexor muscles and fascia because it is believed to not aggravate the spasticity and is widely used in clinical practice. Fascial mobilization will applied regarding the following strategies.

The patient lied on prone position with knee extension and therapist put the patient's plantar surface to her femoral region. Achilles, tibialis posterior, perenous longus and brevis distal tendons, gastrocnemius proximal tendons, hamstring's distal tendons will mobilize at first stage. The second stage of fascia mobilization includes the deep fascial mobilization of posterior crural muscle trunks. After that, the skin also gently mobilize. During fascial mobilization, once the spastic muscles relaxation were appeared, the ankle is been moved to dorsiflexion gradually. FM will carry out for 15 minutes for each foot.

Same patients will receive also stretching exercises consisted of 30 s stretching and 10 s resting periods and will carry out for 15 minutes for each foot at second day after the first evaluation.Fourteen healthy volunteers will receive no interventions.

Assessments will utilize at initially and after FM were applied at first visit. The day after patients will asked to come again and initially evaluations will repeat before stretching exercises. After stretching exercises patients will evaluate again with same tools.

Assessment tools described as following: Modified Ashworth scale will use to evaluate of severity of plantar flexor spasticity. Static and dynamic loading parameters will be evaluate with pedobarography.Maximum loading pressure -N/cm2, maximum loading time- ms for; 1st. and 5th metatarsal head, medial and lateral heel and midfoot will be recorded both while the patients standing and walking.

ELIGIBILITY:
Inclusion Criteria:

* Want to participate
* Individuals with multiple sclerosis who can walk alone for 50 meters
* Healthy participants who diagnosed no disorders or orthopedic problems.

Exclusion Criteria:

* Do not want to participate
* Surgery history

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pedobarography for assessment of foot pressure while standing and walking. | Initially evaluation at first minute, Change from initial evaluation to 20th minutes, Change from initial evaluation to 24 hours, Change from initial evaluation to 24 hours and 20 minutes
  Participant stands and walks on system name is pedobarography which records foot pressure, for 7 minutes. Foot pressure means, gravitational force reflecting from ground at every foot step phase. Newton/cm2 is the unit of measure.

SECONDARY OUTCOMES:
Modified Ashworth Scale for evaluation of severity of involuntary muscle contraction | Initially evaluation at first minute, at 20th minutes, at 24 hours, at 24 hours and 20 minutes
  Modified Ashworth Scale is an assessment method gives severity of involuntary contraction of muscle. Evaluator gives point from 0 to 4 according to muscle reflection to stretching